CLINICAL TRIAL: NCT01880346
Title: Vehicles for the Absorption of Vitamin D in Cystic Fibrosis: Comparison of Powder vs Oil
Brief Title: Comparison of Absorption of Vitamin D in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, MD, PH.D, Associate Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00066261; Hermes vitamin D (Other: Tangpricha)
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Vitamin D; absorption; vitamin Deficiency; fat soluble
MeSH Terms: conditions — Cystic Fibrosis; Avitaminosis | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100,000 IU D-50 powder (Active Comparator): Vitamin D oil vs powder. 100,000 IU powder form of vitamin D, assessment of D3 absorption. One Dose of vitamin D powder format administered. Absorption rate monitored over 72 hour period
  Interventions: Dietary Supplement: Vitamin D Powder
- 100,000 IU Maximum D3 in oil (Active Comparator): Vitamin D oil vs powder. One Dose of 100,000 IU vitamin D oil format administered. Absorption rate monitored over 72 hour period
  Interventions: Dietary Supplement: Vitamin D Oil

INTERVENTIONS:
Dietary Supplement: Vitamin D Powder — Patients will be randomly assigned to a powder supplement of 100,000 IU vitamin D3. Randomization will be in blocks of 4 (meaning for every 4 subjects there will be 2 vitamin D and 2 placebo treated patients). Blood will be drawn by IV catheter at baseline, 2, 4, 8, 12, 24, 48, and 72 hours after vitamin D3 dosing
  Other Names: D3-50 Cholecalciferol
  Arms: 100,000 IU D-50 powder
Dietary Supplement: Vitamin D Oil — Patients will be randomly assigned to an oil based supplement of 100,000 IU vitamin D3. Randomization will be in blocks of 4 (meaning for every 4 subjects there will be 2 vitamin D and 2 placebo treated patients). Blood will be drawn by IV catheter at baseline, 2, 4, 8, 12, 24, 48, and 72 hours after vitamin D3 dosing
  Other Names: Maximum D3
  Arms: 100,000 IU Maximum D3 in oil

SUMMARY:
The investigators predict that a powder pill form of vitamin D will be more effectively absorbed than an oil form of vitamin D in people diagnosed with Cystic Fibrosis.

DETAILED DESCRIPTION:
The purpose of this study is to see how well two different forms of vitamin D work in Cystic Fibrosis (CF). Patients with Cystic Fibrosis have a hard time absorbing certain foods and often have low vitamin D levels. Studies show that vitamin D may help fight infections common in Cystic Fibrosis. The investigators would like to see if a powder pill form of vitamin D will work better than a pill mixed with oil. Each person will randomly receive either a powder pill or an oil based pill. Blood will be tested while during a 3-4 day hospital stay. The investigators plan to enroll no more than 24 patients with CF from Emory University Hospital for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult CF patients (age >18 years
* Able to tolerate oral medication
* Expected to survive the duration of the study

Exclusion Criteria:

* Inability to obtain or declined informed consent from the subject and/or legally authorized representative
* History of disorders associated with hypercalcemia
* Current hypercalcemia (albumin-corrected serum calcium >10.8 mg/dL or ionized calcium >5.2 mg/dL)
* Chronic kidney disease worse than stage III (<60 ml/min), 7) Forced Expiratory Volume (FEV1)% predicted <20%
* Current significant hepatic dysfunction total bilirubin > 2.5 mg/dL with direct bilirubin > 1.0 mg/dL
* Current use of cytotoxic or immunosuppressive drugs
* History of AIDS or illicit drug abuse
* too ill to participate in study based on investigator's or study team's opinion
* current enrollment in another intervention trial

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of Absorption of vitamin D3 to blood | 72 hours
  rates of absorption of D3 will be compared for either an oil based or powder form pill OVER 72 HOURS.

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Grossmann RE, Zughaier SM, Liu S, Lyles RH, Tangpricha V. Impact of vitamin D supplementation on markers of inflammation in adults with cystic fibrosis hospitalized for a pulmonary exacerbation. Eur J Clin Nutr. 2012 Sep;66(9):1072-4. doi: 10.1038/ejcn.2012.82. Epub 2012 Jul 18. PMID 22805498
- [Result] Tangpricha V, Kelly A, Stephenson A, Maguiness K, Enders J, Robinson KA, Marshall BC, Borowitz D; Cystic Fibrosis Foundation Vitamin D Evidence-Based Review Committee. An update on the screening, diagnosis, management, and treatment of vitamin D deficiency in individuals with cystic fibrosis: evidence-based recommendations from the Cystic Fibrosis Foundation. J Clin Endocrinol Metab. 2012 Apr;97(4):1082-93. doi: 10.1210/jc.2011-3050. Epub 2012 Mar 7. PMID 22399505
- [Result] Tangpricha V, Koutkia P, Rieke SM, Chen TC, Perez AA, Holick MF. Fortification of orange juice with vitamin D: a novel approach for enhancing vitamin D nutritional health. Am J Clin Nutr. 2003 Jun;77(6):1478-83. doi: 10.1093/ajcn/77.6.1478. PMID 12791627
- [Result] Johnson EJ, Krasinski SD, Howard LJ, Alger SA, Dutta SK, Russell RM. Evaluation of vitamin A absorption by using oil-soluble and water-miscible vitamin A preparations in normal adults and in patients with gastrointestinal disease. Am J Clin Nutr. 1992 Apr;55(4):857-64. doi: 10.1093/ajcn/55.4.857. PMID 1550069
- [Result] Roum JH, Buhl R, McElvaney NG, Borok Z, Crystal RG. Systemic deficiency of glutathione in cystic fibrosis. J Appl Physiol (1985). 1993 Dec;75(6):2419-24. doi: 10.1152/jappl.1993.75.6.2419. PMID 8125859
- [Result] Hecker TM, Aris RM. Management of osteoporosis in adults with cystic fibrosis. Drugs. 2004;64(2):133-47. doi: 10.2165/00003495-200464020-00002. PMID 14717616
- [Derived] Hermes WA, Alvarez JA, Lee MJ, Chesdachai S, Lodin D, Horst R, Tangpricha V. Prospective, Randomized, Double-Blind, Parallel-Group, Comparative Effectiveness Clinical Trial Comparing a Powder Vehicle Compound of Vitamin D With an Oil Vehicle Compound in Adults With Cystic Fibrosis. JPEN J Parenter Enteral Nutr. 2017 Aug;41(6):952-958. doi: 10.1177/0148607116629673. Epub 2016 Feb 22. PMID 26903303